CLINICAL TRIAL: NCT00166374
Title: Outcomes Following Balloon Kyphoplasty for Vertebral Compression Fracture
Brief Title: To Evaluate Success of Cement Treatment of Spinal Compression Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1707-05
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Kyphoplasty

INTERVENTIONS:
Procedure: balloon kyphoplasty

SUMMARY:
Patients with vertebral compression fracture will be treated cement injection into the spine and monitored using standard evaluations.

DETAILED DESCRIPTION:
Patients with vertebral compression fracture will be diagnosed and treated with balloon kyphoplasty. Pain and functional status will be assessed at baseline, 1-, 12-, and 24-months post-operatively using VAS pain scale, Oswestry Disability Index, and SF-36.

ELIGIBILITY:
vertebral compression fracture

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
pain
disability

CONTACTS AND LOCATIONS:
Overall Officials: H. Gordon Deen, Jr., M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States